CLINICAL TRIAL: NCT00335140
Title: Phase II Study of Rituximab Given in Conjunction With Standard Chemotherapy in Primary Central Nervous System (CNS) Lymphoma
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Primary Central Nervous System Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000475776; ECOG-E1F05 (Other: ECOG-ACRIN)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Cytarabine; Dexamethasone; Calcium Dobesilate; dexamethasone 21-phosphate; dexamethasone acetate; Leucovorin; Methotrexate; Procarbazine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab + standard chemotherapy (Experimental): Rituximab + high dose methotrexate, leucovorin, vincristine, procarbazine, dexamethasone, and cytarabine. Patients with meningeal involvement will receive additional methotrexate and leucovorin.
  Interventions: Biological: Rituximab; Drug: Cytarabine; Drug: Dexamethasone; Drug: Leucovorin; Drug: Methotrexate; Drug: Procarbazine; Drug: Vincristine

INTERVENTIONS:
Biological: Rituximab — Rituximab is administered intravenously. The initial rate is 50 mg/hr for the first hour. If no toxicity is seen, the rate may be escalated gradually in 50 mg/hour increments at 30-minute intervals to a maximum of 300 mg/hr. If the first dose is well tolerated, the initial rate for subsequent dose is 100 mg/hr, increased gradually in 100 mg/hr increments at 30-minute intervals, not to exceed 400 mg/hr.
  Other Names: Rituxan
Drug: Cytarabine — 3 g/m2/day in 500 cc D5W IV over 2 hrs. x 2 doses 24hrs. apart, Weeks 11, 14
  Other Names: Cytosar-U; Ara-C; Arabinosylcytosine
Drug: Dexamethasone — 16mg (week 1) PO daily Weeks 1, 2, 3, 4, 5, 6 Taper by 4 mg/wk, weeks 2, 3, by 2 mg/wk week 4, 5, 6
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex; dexamethasone sodium phosphate; dexamethasone acetate
Drug: Leucovorin — 25 mg PO/IV every 6 hrs. x 12 doses, Weeks 1, 3, 5, 7, 9 For patients with meningeal involvement additionally 10 mg PO every 12 hrs. x 8 doses, Weeks 2, 4, 6, 8, 10
  Other Names: leucovorin calcium
Drug: Methotrexate — 3.5 g/m2In 500 cc D5W + 25 mEq NaHCO3 IV over 2 hours, Weeks 1, 3, 5, 7, 9
  For patients with meningeal involvement additionally:
  12 mg Intrathecally, in preservative-free sterile .9NS Weeks 2, 4, 6, 8, 10 Via Ommaya or lumbar puncture
  Other Names: Otrexup; Rasuvo; Rheumatrex; Trexall; Amethopterin; Methotrexate Sodium; MTX
Drug: Procarbazine — 100 mg/m2 PO daily x 7 days Weeks 1, 5, 9
  Other Names: Matulane; Procarbazine hydrochloride
Drug: Vincristine — 1.4 mg/m2 IV push, Weeks 1, 3, 5, 7, 9 2m2 (2.8 mg) dose cap
  Other Names: Vincristine Sulfate; Oncovin; Vincasar; LCR; VCR

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as methotrexate, leucovorin, vincristine, procarbazine, dexamethasone, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy works in treating patients with primary central nervous system (CNS) lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate.

Secondary

* Determine the progression-free survival of these patients.
* Determine the proportion of progression-free and overall survival in these patients.
* Determine rituximab cerebrospinal fluid pharmacokinetics (only in patients requiring intrathecal chemotherapy).

OUTLINE: This is a multicenter study.

Patients receive rituximab IV 3 times weekly in weeks 1-4; high-dose methotrexate IV over 2 hours in weeks 1, 3, 5, and 9; oral or IV leucovorin calcium every 6 hours for 12 doses beginning 24 hours after the start of methotrexate in weeks 1, 3, 5, and 9; vincristine IV in weeks 1, 3, 5, 7, and 9; oral procarbazine hydrochloride daily on days 1-7 in weeks 1, 5, and 9; oral dexamethasone daily in weeks 1-6; and cytarabine IV over 2 hours twice weekly in weeks 11 and 14.

Patients with positive cerebrospinal fluid also receive methotrexate intrathecally and oral leucovorin calcium every 12 hours for 8 doses beginning 24 hours after the start of methotrexate in weeks 2, 4, 6, 8, and 10.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed non-Hodgkin's lymphoma by brain biopsy
* Patients with inconclusive biopsy or patients who are not candidates for biopsy must have typical CT scan or MRI of the brain AND meet ≥ 1 of the following criteria:

  * Positive cerebrospinal fluid cytology for lymphoma OR a monoclonal lymphoid population as defined by cell surface markers or immunoglobulin gene rearrangement studies
  * Biopsy-proven involvement of the vitreous or uvea if cells are apparent in the posterior chamber or vitreous by ophthalmological examination
* Bideminsionally measurable disease, defined as contrast-enhancing tumor ≥ 1 cm by pretreatment MRI/CT scan

  * Meningeal or vitreous involvement constitutes evaluable but not measurable disease
  * If an excisional, rather than a needle biopsy was done, measurable disease must be present on a postoperative scan (not a PET-CT scan)
* ECOG performance status 0-3
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ upper limit of normal (ULN)
* SGOT ≤ 2.0 times ULN
* Creatinine clearance ≥ 50 mL/min
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Pregnant or nursing
* HIV-1 positivity
* Other malignancy within the past 5 years except basal cell skin cancer or any carcinoma in situ
* Pre-existing immunodeficiency
* Hepatitis B surface antigen positivity
* Systemic lymphoma (as determined by pre-registration CT scans and physical examination)
* Prior chemotherapy or radiotherapy for primary central nervous system lymphoma
* Prior organ or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-08-23 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lode J. Swinnen, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Deborah T. Blumenthal, MD, Study Chair — University of Utah
Locations (68):
- United States (68):
  - Stanford Cancer Center, Stanford, California
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Derived] Swinnen LJ, O'Neill A, Imus PH, Gujar S, Schiff D, Kleinberg LR, Advani RH, Dunbar EM, Moore D, Grossman SA. Phase II study of rituximab given in conjunction with standard chemotherapy in primary central nervous system lymphoma (PCNSL): a trial of the ECOG-ACRIN cancer research group (E1F05). Oncotarget. 2017 Nov 6;9(1):766-773. doi: 10.18632/oncotarget.22332. eCollection 2018 Jan 2. PMID 29416652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG-ACRIN member institutions starting 12/21/2006 and accrued its first patient on 08/23/2007. The study was suspended 2/24/2010 for interim analysis. After the interim analysis, it was determined that the goals of the study had been met and the study was closed on 4/12/2013.
Groups:
- Rituximab + Standard Chemotherapy: rituximab
  cytarabine
  dexamethasone
  leucovorin calcium
  methotrexate
  procarbazine hydrochloride
  vincristine sulfate
Period: Overall Study
Arm/Group | Rituximab + Standard Chemotherapy
Started | 26
Eligible | 25
Treated | 25
Completed | 25
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy
Arm/Group | Rituximab + Standard Chemotherapy
Number analyzed (Participants) | 25
Age, Customized [Count of Participants; unit: Participants] — Older or younger than 60
  Participants
    Age: Age < 60 years | 15
    Age: Age ≥ 60 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 24
  Race: Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 25
ECOG Performance Status [Count of Participants; unit: Participants] — 0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  Participants
    0 | 1
    1 | 15
    2 | 5
    3 | 4
Neurologic Function Status [Count of Participants; unit: Participants]
  No symptoms | 0
  Minor symptoms | 11
  Moderate symptoms/fully active | 5
  Moderate symptoms/less than fully active | 7
  Severe neurologic symptoms | 2
Cerebrovascular Disease [Count of Participants; unit: Participants]
  Never | 21
  Symptomatic or on medication | 4
Other Medical Problems at Baseline [Count of Participants; unit: Participants]
  Never | 9
  Symptomatic or on medication | 7
  Past history of | 7
  Missing/unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate - Locally Reviewed
Description: Assessed by the ECOG-ACRIN data manager based upon local review of images and data sent by the local sites.
  Treatment response was determined by calculating the sum of the maximal cross section in 2 separate axes using enhancing lesion(s) on CT or MRI imaging. The same imaging modality was to be used throughout assessment. Complete response was defined as the disappearance of all contrast enhancing tumor size on CT or MRI, patient was off all glucocorticoids, and resolution of all meningeal and vitreous involvement if present. Response must have lasted at least 4 weeks.
Time Frame: For the primary endpoint, complete response will be based on disease status at three weeks post the end of therapy (week 17).
Population: Eligible, treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Standard Chemotherapy
Number analyzed (Participants) | 25
percentage of participants | 64 [42.5 to 82]

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks during treatment and once for the 30 days following the last dose of protocol drug, or until the initiation of subsequent treatment, whichever comes first.
Arm/Group | Rituximab + Standard Chemotherapy
Serious Adverse Events (participants affected / at risk) | 24/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Standard Chemotherapy (N=26)
Anemia (Blood and lymphatic system disorders) | 6
Leukocytes decreased (Investigations) | 17
Lymphopenia (Investigations) | 10
Neutrophils decreased (Investigations) | 20
Platelets decreased (Investigations) | 5
Fatigue (General disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Muco/stomatitis (symptom) esophagus (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Perforation, colon (Gastrointestinal disorders) | 1
Perforation, stomach (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Infection Gr0-2 neut, upper aerodig (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 2
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Neuropathy CN VI lateral deviation eye (Nervous system disorders) | 1
Neuropathy-motor (Nervous system disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 3
Esophagus, pain (Gastrointestinal disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Head/headache (Nervous system disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Oral cavity, pain (Gastrointestinal disorders) | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Standard Chemotherapy (N=26)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Anemia (Blood and lymphatic system disorders) | 23
Leukocytes decreased (Investigations) | 24
Lymphopenia (Investigations) | 12
Neutrophils decreased (Investigations) | 11
Platelets decreased (Investigations) | 19
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 5
Fatigue (General disorders) | 21
Insomnia (Psychiatric disorders) | 6
Rigors/chills (General disorders) | 4
Weight gain (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Wound - non-infectious (Injury, poisoning and procedural complications) | 2
Anorexia (Metabolism and nutrition disorders) | 6
Constipation (Gastrointestinal disorders) | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 13
Taste disturbance (Nervous system disorders) | 4
Vomiting (Gastrointestinal disorders) | 7
Petechiae (Skin and subcutaneous tissue disorders) | 2
Edema limb (General disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Alkaline phosphatase increased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 15
Aspartate aminotransferase increased (Investigations) | 11
Acidosis (Metabolism and nutrition disorders) | 2
Blood bilirubin increased (Investigations) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 15
Creatinine increased (Investigations) | 13
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 16
Hyponatremia (Metabolism and nutrition disorders) | 13
Metabolic/Laboratory-other (Investigations) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Extremity-lower (gait/walking) (General disorders) | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 4
Neuropathy-motor (Nervous system disorders) | 5
Neuropathy-sensory (Nervous system disorders) | 10
Personality (Psychiatric disorders) | 2
Speech impairment (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Vision-blurred (Eye disorders) | 3
Tearing (Eye disorders) | 2
Abdomen, pain (Gastrointestinal disorders) | 2
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2
Head/headache (Nervous system disorders) | 7
Muscle, pain (Musculoskeletal and connective tissue disorders) | 6
Oral cavity, pain (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Urinary frequency/urgency (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No